CLINICAL TRIAL: NCT04294082
Title: Evaluating a Brief Mindfulness-based Intervention for Parents of Adults With Intellectual Disabilities: a Case Series.
Brief Title: Study of Mindfulness Course for Parents of Adults With Intellectual Disabilities
Status: Withdrawn | Type: Observational
Why Stopped: Study stopped due to the outbreak of the covid-19 pandemic.
Sponsor: University of Edinburgh (Other)
Collaborators: NHS Grampian (Other Government)
Responsible Party: Sponsor
Other Study IDs: CAHSS1912/05
Record Dates: First submitted 2020-02-21; First posted 2020-03-03 (Actual); Last update posted 2020-08-21 (Actual); Status verified 2020-03

CONDITIONS: Intellectual Disability
MeSH Terms: conditions — Intellectual Disability

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Mindfulness based intervention: A shortened version of a mindfulness-based intervention originally developed by Jon Kabat-Zinn for management of chronic pain.
  Interventions: Behavioral: Mindfulness based intervention

INTERVENTIONS:
Behavioral: Mindfulness based intervention — A four session, 120 mins per session mindfulness based course delivered weekly oer the course of four weeks. The mindfulness sessions are based on the model delineated by Kabat-Zinn (1992) and will encompass:
  * an introduction to mindfulness
  * body-scan exercises
  * sitting meditation
  * mindful movement exercises
  * individual and group reflections
  * homework exercises

SUMMARY:
Being a parent to an adult person with learning disabilities can be very stressful, and can lead to experiencing mental health problems. Not much is known about what sort of support services should be offering to these parents; and not many options are available as a result. This study will try to find out if a short intervention, known as a mindfulness-based intervention (MBI), can be of help to these families. A mindfulness-based intervention is one that aims to increase someone's mindfulness, which is the ability to be aware of the present, in a non-judgemental fashion.

Simply put, what the investigators would like to find out from this study is: "Can a short course of MBI help improve the well-being of parents of adults with learning disabilities?"

To answer this question, the investigators will seek to invite parents to attend a mindfulness course of the duration of 4 sessions. Parents will be invited to participate by NHS staff at their local Community Learning Disabilities Team, who will hand out information sheets and consent forms. Parents will be informed that they may choose to withdraw from the study at any time without this having any negative effect. The investigators will also ask parents to provide feedback on their experience of the course using online questionnaires. Parents will be asked to complete the questionnaires at 6 points: 1 month before the start of the course, at the start of the course, at the end of the course, and at 3, 6 and 12 months after the course has ended. This way, the investigators will be able to track any changes in how parents rate their well-being; and if these changes persist in the long-term.

At the end of the study, participants will be offered information on the results.

DETAILED DESCRIPTION:
A multitude of studies has established that parenting a child with intellectual disabilities (IDs) can negatively influence the psychological and physical wellbeing of primary caregivers. The same correlation between IDs and parental psychological distress exists in the parents of adults with IDs, with the transition from childhood to adulthood being particularly detrimental to the psychological wellbeing of the family. Carers of children with IDs often report increased levels of parental stress, a feature that is amplified in some categories of IDs, such as in autism spectrum disorder. Importantly, the effects of this especially demanding relationship are not limited to impacting the carers' wellbeing alone; they can also affect the carers' ability to respond to problematic child behaviour, and result in financial hardship.

In terms of psychological distress on the part of people with intellectual disabilities (PWIDs), this is most often observed in the form of challenging behaviour, which can be used by PWIDs to communicate their distress. Of interest to the present study, the complex and enduring pattern of difficulties observed within these families cannot be accounted for purely by the psychological distress of the carers, nor does it stem from challenging behaviour alone. Instead, it has been proposed that the relationship between parental stress and the child's challenging behaviour is bi-directional, and self-reinforcing, in that parental stress can increase challenging behaviour, just as challenging behaviour can induce stress, and other forms of psychological distress. This pattern has been observed in families with children, as well as in families with adults with IDs.

Given the link between challenging behaviour, parental stress, and their interdependent nature, there has recently been a focus on employing therapeutic modalities that are explicitly aimed at reducing stress, with third-wave cognitive behavioural therapies (CBT) at the forefront of such scrutiny. Among third-wave CBTs, mindfulness-based interventions (MBIs) have been employed with especially promising results, making them veritable candidates as effective interventions for what is a sizeable segment of the population.

MBI adaptations

It should be noted that the increased range of applicability derived from said universality can limit the scope and clarity of the MBIs' research base. Specifically, as observed in a recent review on the efficacy of MBIs in parents of children with disabilities, a plethora of different interventions and adaptations of MBIs are continuously being developed, from the classic programmes devised by Jon Kabat-Zinn and his team, to hybrid interventions that combine MBIs with other therapies, such as DBT or ACT. Such abundance of variation can limit the precision with which the various MBIs are comparable with one another, and frustrates the search for a definite analysis of precisely which mindfulness factors contribute to the self-reported decreases in psychological distress. In parallel, efforts are being made to distil the essential criteria a mindfulness intervention should be based on.

MBIs can also be adapted in relation to their structure, not just by intervention modality they incorporate. Shortened versions of MBIs have been devised and tested with positive results, with effect sizes for psychological outcomes comparable to those found in programmes of classic length. Shortened MBIs can cover the same content as their lengthier counterparts, within fewer sessions; or they may simply reduce the content they cover, and provide that within fewer sessions. In both instances, the literature suggests that there is no significant correlation between psychological outcomes and course length, indicating that shortened versions of MBIs may achieve the same psychological outcomes by the end of the programme, in clinical, as well as non-clinical populations.

Presently, no robust research exists on what intervention works best for parents of PWIDs, particularly within the realm of adults with IDs. To the author's knowledge, only one study has to date explored the effectiveness of a short MBI aimed specifically at parents of adults with a disability. It should be noted, however, that the study primarily evaluated parents of adults with a diagnosis of autism spectrum disorder (ASD). This limits the generalisability of the study to the ASD population, which represents but a section of the population with IDs. In addition, the authors of the study acknowledge that parents of adult children with IDs often find it difficult to commit to a course of MBI due to the time constrains dictated by their children's needs, and recommend the trialling of even shorter MBIs, with no studies to date having evaluated an MBI as brief as the one proposed herein. Finally, despite there being extensive research on the shorter-term effects of MBIs, no study to date has focussed with sufficient emphasis on the longer-term effects of MBI course. Advancing our understanding of whether MBIs retain their effect over time can lead to substantial improvements in terms of clinical applications.

Based on the premises that:

1. shortened versions of MBIs have successfully generated psychological change in comparable populations; and
2. theoretical models relating to children with disabilities suggest that parental stress negatively influences the caregiver-offspring dyad;

it is hypothesized that a 4-week MBI course will achieve positive psychological outcomes in this population.

ELIGIBILITY:
Inclusion Criteria:

* All parents of adults (defined as individuals aged 16 years or above) with IDs, identified by the CLDT will be eligible.
* No formal diagnosis of IDs will be sought, as often service users do not have a formal diagnosis due to a lack of diagnostic services being available (either historically, or presently).

Exclusion Criteria:

* Parents of children (under 16 years old) with IDs. This includes family units comprised of both children and adults with IDs.
* Parents who are not sufficiently fluent in English, or who themselves have an IDs, such that they might be unable to undertake the intervention and complete the relative outcome measures.
* Parents that do not have capacity to consent to research at the time it is sought.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Parents of adults with IDs living in Aberdeenshire.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2020-04-01 (Estimated); Primary Completion 2021-10-01 (Estimated); Study Completion 2021-10-01 (Estimated)

PRIMARY OUTCOMES:
Parental Stress Scale | Baseline (4 weeks before the start of the mindfulness course); Pre- (at the start of the mindfulness course); Post- (at the end of the mindfulness course; Time point: 4 weeks); Follow-ups (at 3, 6, 12 months from the end of the mindfulness course)
  Self-reported questionnaire measuring change in levels of stress in parents. Scores on scale range from 1 to 5, with higher values indicating lower parental stress.

SECONDARY OUTCOMES:
Warwick-Edinburgh Mental Well-Being Scale | Baseline (4 weeks before the start of the mindfulness course); Pre- (at the start of the mindfulness course); Post- (at the end of the mindfulness course; Time point: 4 weeks); Follow-ups (at 3, 6, 12 months from the end of the mindfulness course)
  Self-reported questionnaire measuring changes in psychological well-being. Scores on scale range from 1 to 5, with higher values indicating higher levels of well-being.
Five-facet Mindfulness Questionnaire, Short Form. Scores on each questionnaire item range from 1 to 5, with higher values indicating higher levels of mindfulness. | Baseline (4 weeks before the start of the mindfulness course); Pre- (at the start of the mindfulness course); Post- (at the end of the mindfulness course; Time point: 4 weeks); Follow-ups (at 3, 6, 12 months from the end of the mindfulness course)
  Self-reported questionnaire measuring changes in levels of mindfulness
Satisfaction with Life Scale. Scores range from 1 to 7, with a higher score indicating higher satisfaction with life. | Baseline (4 weeks before the start of the mindfulness course); Pre- (at the start of the mindfulness course); Post- (at the end of the mindfulness course; Time point: 4 weeks); Follow-ups (at 3, 6, 12 months from the end of the mindfulness course)
  Self-reported questionnaire measuring changes in satisfaction with life

CONTACTS AND LOCATIONS:
Overall Officials: Matteo Turco de Pretis-Cagnodo, MSc, Principal Investigator — University of Edinburgh

IPD SHARING:
Plan to Share IPD: No